CLINICAL TRIAL: NCT02922608
Title: French National Investigation About Student's Sleep Perturbations Before Simulation Session.
Brief Title: French Survey About Student's Sleep Perturbations Before Simulation Session.
Acronym: Simsleep
Status: Completed | Type: Observational
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Lilot Marc, MD, Claude Bernard University
Other Study IDs: simusleepsurvey
Record Dates: First submitted 2016-09-30; First posted 2016-10-04 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Sleep; Anxiety
Keywords: Education, Medical
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: simulation practice — simulation session

SUMMARY:
High fidelity simulation provide educational skills but the simulation of critical events could eventually provide anxiety among participants.

The anxiety could raise before the simulation session and affect the perceived quality of sleep the night prior to the simulation session. The lack of sleep would eventually affect both participation and memorization during the simulation session. The investigators would like to investigate with a survey how much participants had their sleep affected before the simulation session.

DETAILED DESCRIPTION:
High fidelity simulation provide educational skills but the simulation of critical events could eventually provide anxiety among participants.

The anxiety could raise before the simulation session and affect the perceived quality of sleep the night prior to the simulation session. The lack of sleep would eventually affect both participation and memorization during the simulation session.

The investigators would like to investigate with a survey how much participants had their quantity and quality of sleep affected before the simulation session.

ELIGIBILITY:
Inclusion Criteria:

* french talking residents coming to high fidelity simulation

Exclusion Criteria:

* refusal to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: residents coming to simulation center for high fidelity simulation education program.
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Actual)
Dates: Start 2016-10; Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
modification of the sleeping Leeds test | day 1

SECONDARY OUTCOMES:
incidence of sleep perturbations | day 1
analysis of demographics and sleep perturbations | day 1

CONTACTS AND LOCATIONS:
Overall Officials: jean-jacques lehot, PHD, Study Chair — Cless
Locations (1):
- CLESS, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: Undecided